CLINICAL TRIAL: NCT05084729
Title: A Multi-Center InternatiONal Registry to Evaluate the Efficacy oF Imaging With Opto-acoustics to Diagnose BrEast CaNCEr
Brief Title: CONFIDENCE Registry
Acronym: CONFIDENCE
Status: Completed | Type: Observational
Sponsor: Seno Medical Instruments Inc. (Industry)
Collaborators: American College of Radiology (Other)
Responsible Party: Sponsor
Other Study IDs: CONFIDENCE-01
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-01

CONDITIONS: Breast Abnormality Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Imagio OA/US: Imagio optoacoustic
  Interventions: Device: Imagio OA/US

INTERVENTIONS:
Device: Imagio OA/US — Imagio optoacoustic

SUMMARY:
This registry has been designed to obtain real-life, post-market data on the use of the Imagio breast imaging system. This registry is sponsored by Seno Medical Instruments, Inc., the manufacturer of the device.

DETAILED DESCRIPTION:
This is a prospective, controlled, multi-center, observational international registry designed to evaluate the Imagio breast imaging system. The registry will be conducted at up to 12 international centers. Investigators will use Imagio US (IUS) and/or Imagio OA/US imaging per standard of care, anddata will be collected accordingly. Additional imaging and biopsy/surgery will be conducted per standard of care to reach a final diagnosis.

ELIGIBILITY:
Inclusion Criteria - Subjects must meet all the following criteria to be included in the registry:

1. Have been informed of the nature of the registry and provided written informed consent, prior to initiation of any registry activities,
2. Are females 18 years of age or older at the time of consent,
3. Have been referred for a breast US and are subject to treatment with the Imagio breast imaging system.

Exclusion Criteria - Aligned with the contraindications on the use of the device, subjects who meet any of the following criteria will be excluded from the registry:

1. Are pregnant.
2. Have open sores including insect bites, rash, poison ivy, and chafing on the skin of the ipsilateral breast.
3. Are experiencing photo-toxicity associated with currently taking, or having taken, photosensitizing agents within the previous 72 hours such as sulfa, ampicillin, tetracycline.
4. Are currently undergoing phototherapy.
5. Have a history of any photosensitive disease (e.g., porphyria, lupus erythematosus).
6. Are undergoing treatment for a photosensitive disease and is experiencing photosensitivity.
7. Have previously participated in this registry,
8. Are currently enrolled in another investigational study or registry that would directly interfere with the current registry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of up to 600 subjects will be enrolled in the registry in up to 12 sites in the EU and US, with a maximum of 50-100 subjects per site.
  Subjects with lesions/masses presenting with BI-RADS 0-6 will be enrolled. Enrollment into the registry will allow for only 100 lesions/masses presenting with BI-RADS 1 and 2 breast imaging findings and evaluated with the Imagio breast imaging system and 50 lesions/masses presenting with BI-RADS 0 findings and evaluated with the Imagio breast imaging system. This limitation is applicable in order to ensure a cross section of BI-RADS categories enrolled in the registry.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Specificity, negative likelihood ratio, sensitivity and positive likelihood | September 2024
  This parameter will be reviewed for the Intention-to-Diagnose (ITD) and Per-Protocol (PP) populations
Assessment of the percentage of masses that the Imagio system alone or in combination with other imaging modalities is indicated as impacting the decision to biopsy | September 2024
  This parameter will be reviewed for the Intention-to-Diagnose (ITD) and Per-Protocol (PP) populations
Quality of Life Assessment - Testing Morbidity Index | September 2024
  This parameter will be reviewed for the Intention-to-Diagnose (ITD) and Per-Protocol (PP) populations
In malignant breast masses, to assess the roles of the Imagio OA/US as a prognostic biomarker | September 2024
  i.e., the correlation of Imagio OA/US feature scoring with histologic grade, ER and PR hormone receptors, HER2 receptor (IHC and/or HER2 FISH), Ki-67 proliferative index, as well as with molecular subtypes of breast cancer.
  This parameter will be reviewed for the Intention-to-Diagnose (ITD) and Per-Protocol (PP) populations

SECONDARY OUTCOMES:
Characteristics of lymph node lesions/masses the device is used for | September 2024
  This parameter will be reviewed for the Safety population
Incidence and nature of device deficiencies (i.e. device complaints, device malfunctions) | September 2024
  This parameter will be reviewed for the Safety population
Incidence and nature of device and procedure related adverse events | September 2024
  This parameter will be reviewed for the Safety population

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - University Medical Center Groningen, Groningen
  - Zorggroep Twente, Hengelo

IPD SHARING:
Plan to Share IPD: Yes
Your medical history, information from your medical record (i.e., Imagio images, other standard imaging (screening/diagnostic ultrasounds, MRI, diagnostic ultrasound, Mammography, etc.), pathology results, and other information you give us during an interview or from questionnaires, demographic information like your age, ethnicity or race). In an effort to protect your privacy, the study staff will use code numbers instead of your name, to identify your health information. Initials and numbers will be used on any photocopies of your study records. If the results of this study are reported in medical journals or at meetings, you will not be identified. Every effort is made to ensure that your personal information is removed from these images.
Supporting Information: CSR
Time Frame: September 2024
Access Criteria: The following groups can access the IPD.
  To assess accuracy of Imagio:
  * Study staff
  * Imaging Core Lab
  * Seno
  * Doctors, independent of your doctor's office
  Institutions and other persons who are required to review research and monitor medical products/therapies and the conduct of research:
  * FDA
  * DHHS
  * Other U.S. and foreign government authorities
  * Institutional Review Boards
  * Seno representatives